CLINICAL TRIAL: NCT06550882
Title: Post-Marketing Surveillance (Use-result Surveillance) of OBIZUR Injection [Susoctocog Alpha (Porcine Antihemophilic Factor VIII, Recombinant)] for the Approved Indications in South Korea
Brief Title: A Study of OBIZUR in Adults With Acquired Hemophilia A (AHA) in South Korea
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-672-4002
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acquired Hemophilia A
Keywords: Drug Therapy
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- All Participants: Participants with AHA who are receiving OBIZUR injection or initiate OBIZUR Injection treatment for the first time will be enrolled. Both retrospective and prospective participants data will be collected. Retrospective data will be collected from the date of first treatment with OBIZUR injection after the marketing authorization in Korea but before date of signed informed consent and prospective data will be collected from the date of signed informed consent. The treatment and follow up of the participants will be determined by the treating physicians according to her/his routine practice.
  Interventions: Drug: OBIZUR

INTERVENTIONS:
Drug: OBIZUR — OBIZUR injection.
  Other Names: Susoctocog Alpha; Porcine Antihemophilic factor VIII, Recombinant; TAK-672

SUMMARY:
Acquired hemophilia A (AHA) is a rare bleeding condition which prevents blood clotting. Acquired means that people are not born with this condition or have a family history of blood clotting conditions. People living with AHA can have sudden and severe bleeding. They also have longer bleeding compared to people without AHA.

The main aim of the study is to learn how safe OBIZUR is in adults with AHA.

Other aims are to see how effective OBIZUR is to control bleeding and how treatment is used in a routine clinical practice setting.

The treatment of the participants will be determined by the treating physicians.

During the study, data already existing in the participants' medical record and new data will be collected.

DETAILED DESCRIPTION:
This is a prospective, and retrospective, multicenter, single-arm non-interventional post-marketing surveillance study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with AHA.
* Participants who are determined to have the clinical need to receive Obizur treatment.
* Participants aged 18 years or older at time of initiation of Obizur treatment.
* Participants agreed to participate in the study and voluntarily signed the informed consent.

Exclusion Criteria:

* Participants with hypersensitivity to any of the components of this drug.
* Participants with Congenital Hemophilia A with Inhibitors (CHAWI).
* Participants for whom Obizur treatment is contraindicated as per product label.
* Participants who has participated in another clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving a medicinal product or device during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with AHA who are receiving OBIZUR Injection or initiate OBIZUR Injection treatment for the first time will be enrolled.
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs), Causality to AEs, Serious AEs (SAEs) and AEs of Special Interest (AESI) | Up to 3 months
  Number of participants with AEs, causality to AEs, SAEs and AESI will be reported. The investigator will assess the causal relationship (causality) between the medicinal product and the AE using his/her clinical expertise and judgment.
Number of Participants With Expected/Unexpected AEs and SAEs | Up to 3 months
  Unexpected AE is defined as AE that differs from the information in the product label in nature, severity, specificity, or outcome.
Number of Participants With Adverse Drug Reactions (ADRs), Unexpected ADRs, Serious ADRs, Expected SADRs and Unexpected SADRs | Up to 3 months
  An ADR refers to any undesirable and unintended reaction which occurs during or following the administration of the drug, and in which a causal relationship with the drug cannot be ruled out. In the event that a causal relationship with the drug remains unknown amongst reported adverse events, such reaction shall be considered an adverse drug reaction. Serious ADR means noxious or unintended response to a drug that occurs at any dosage and that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening or results in death. Unexpected ADRs is defined as ADR that differs from the information in the product label in nature, severity, specificity, or outcome.
Number of Participants With Special Situation Report (SSR) | Up to 3 months
  SSR include following events: Pregnancy: any case in which a pregnancy participant is exposed to a Takeda Product or in which a female participant or partner of a male participant becomes pregnant following Takeda product.; Breastfeeding: infant exposure from breast milk; Overdose: all information of any accidental or intentional overdose; Drug abuse, misuse or medication error: all information on medicinal product (MP) abuse, misuse of medication error (potential or actual); Suspected transmission of infectious agent: Suspected (in sense of confirmed or potential) transmission of infectious agent by a MP; Lack of efficacy of Takeda Product; accidental/occupational exposure; Use outside the terms of the marketing authorization, also known as "off-label" and "off-label use"; Use of falsified and counterfeit MP; Drug-drug and drug-food interactions; Inadvertent or accidental exposure with or without an AE; Unintended benefit.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Bleeding Control | Up to 3 months
  Overall Bleeding Control will be determined as either bleeding stopped or did not stop.
Time to Achieve Bleeding Control With OBIZUR Injection | Up to 3 months
  Time to achieve bleeding control will be assessed from initiation of OBIZUR Injection (start time) to the time to achieve bleeding control (stop time).
Number of OBIZUR Injection Infusion Required to Achieve Bleeding Control | Up to 3 months
  Number of OBIZUR injection infusion required to achieve bleeding control will be reported.
Dose of OBIZUR Required to Stop the Bleeding | Up to 3 months
  OBIZUR dose required to stop the bleeding will be reported.
Percentage of Participants With Bleeding Events | Up to 3 months
  Bleeding events will be evaluated and reported as re-bleed, concurrent bleed and subsequent bleed. Re-bleed: if it occurs in the same anatomical location and within 72 hours of the resolution of the previous bleeding. Concurrent bleed: if it occurs at the same time (that is, during treatment or within 72 hours of resolution) as previous bleed but at a different anatomical location. Subsequent bleed: if it is a new bleed occurring 72 hours after the resolution of the previous bleed (either in the same anatomical location or in a new one).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/333b153685d74d6b??page=1&idFilter=TAK-672-4002